CLINICAL TRIAL: NCT01180387
Title: Reproductive Medicine Network Biologic Specimen Repository
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Penn State University (Other); University of Colorado, Denver (Other); University of Michigan (Other); University of Pennsylvania (Other); University of Texas (Other); University of Vermont (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Heping Zhang, Principal Investigator, Yale University
Other Study IDs: RMN-Repository; 5U10HD055925 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-12 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — The RMN plans to collect baseline serum samples (5 cc) and DNA for storage and eventual DNA extraction. The whole blood will also be collected by the clinical sites.
  As part of the RMN effort, pregnancies conceived as part of the study protocols are entered into a pregnancy registry if the subjects consent to be part of the registry. Saliva samples from the child conceived as part of the protocols, as well as the parent from whom the DNA was not collected as part of the original protocols will be collected at that time. The newborn's saliva will be collected with up to 5 saliva sponges, the tips of which are cut off and stored using an Oragene® kit. The adults will be asked to provide 2 cc of saliva, which will be stored with the same kits. These saliva samples will be stored at -20°C.
  Two of the RMN studies involve assessing semen parameters. As part of this protocol, we anticipate collecting semen samples from male subjects.
Oversight: Data Monitoring Committee: No

SUMMARY:
The Reproductive Medicine Network (RMN) is a nationwide cooperative network of 7 clinical sites and a data coordination center, and is sponsored in 5 year increments by The Eunice Kennedy Shriver National Institute for Child Health and Human Development (NICHD). The RMN is charged with designing, implementing and publishing high quality clinical research in reproductive medicine. It has been in existence for over 15 years and has performed several seminal clinical trials that have fundamentally changed clinical practice in this field. In addition, many worthy ancillary protocols have been generated and published.

It is this latter fact, as well as the continued interest by investigators both inside and outside the RMN for access to DNA or serum samples from the previously performed trials, that has motivated the present investigators to proactively begin a biologic samples repository from the ongoing and pending RMN clinical trials. Ideally, this repository would allow investigators to seamlessly access trial samples for many years into the future, and thus greatly amplify the use of resources and the impact of the RMN.

ELIGIBILITY:
Inclusion Criteria:

* Any subject of an RMN clinical trial and consents to participate in the repository is eligible for inclusion.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Current patients of the ongoing and future RMN clinical protocols, who consents to participate in this repository.
Sampling Method: Non-Probability Sample
Enrollment: 1640 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subject who accepted participation | 4.2 years

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Nanette Santoro, MD, Study Chair — University of Colorado, Denver; Peter Casson, MD, Principal Investigator — University of Vermont; Michael Diamond, MD, Study Director — Wayne State University; Richard Legro, MD, Study Director — Pennsylvania State University College of Medicine; William Schlaff, MD, Study Director — University of Colorado Denver Health Science Center; Gregory Christman, MD, Study Director — University of Michigan; Christos Coutifaris, MD, Study Director — University of Pennsylvania; Robert Brzyski, MD, PhD, Study Director — The University of Texas Health Science Center at San Antonio; Heping Zhang, PhD, Study Director — Yale University
Locations (15):
- United States (15):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - University of Connecticut, Storrs, Connecticut
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Hackensack University, Hackensack, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University, School of Medicine, Richmond, Virginia